CLINICAL TRIAL: NCT01359982
Title: A Phase I, Open-Label, Multiple Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of RRx-001 in Subjects With Advanced Solid Tumors or Lymphomas For Which There Are No Currently Accepted Curative Therapies
Brief Title: Safety and Pharmacokinetic Study of RRx-001 in Cancer Subjects
Acronym: DINAMIC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRx001-11-01
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-08

CONDITIONS: Malignant Solid Tumor; Lymphomas
Keywords: Advanced Solid Tumors; Lymphomas; Safety; Blood flow; Nitric oxide; Cancer; Dynamic contrast enhanced MRI (DCE-MRI); Contrast Enhanced Ultrasound (CEUS)
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — RRx-001

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RRx-001 (Experimental)
  Interventions: Drug: RRx-001

INTERVENTIONS:
Drug: RRx-001 — Dose level 1 (10 mg/m2)
Drug: RRx-001 — Dose Level 2 (16.7 mg/m2)
Drug: RRx-001 — Dose Level 3 (24.6 mg/m2)
Drug: RRx-001 — Dose Level 4 (33 mg/m2)
Drug: RRx-001 — Dose Level 5 (55.0 mg/m2)
Drug: RRx-001 — Dose Level 6 (83 mg/m2)

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetic profile of RRx-001 for injection in subjects with advanced solid tumors or lymphomas for which there are no currently accepted curative therapies. This study will also conduct an exploratory evaluation of objective tumor response using CT or MRI.

DETAILED DESCRIPTION:
The DINAMIC (DINitroazetidines As Medications In Cancer) trial represents a provascular approach to temporarily change tumor blood flow and oxygenation. Blood supply to most tumors is poor, causing parts of tumors to have a low oxygen content which promotes aggressiveness and metastasis. The DINAMIC trial uses specific imaging techniques (including ultrasound), biopsy, and breath analysis to provide an early assessment of therapeutic activity.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, aged at least 18 years.
* Subject has a histologically or cytologically confirmed diagnosis of an advanced, malignant, incurable solid tumor(s) or lymphoma that is metastatic and/or unresectable and/or for which standard curative measures either are not applicable, or do not exist, or are no longer effective. Subjects with curative treatment options are not eligible for the protocol.
* Subject is not receiving any active treatment for his/her malignancy (except for prostate cancer subjects receiving luteinizing hormone-releasing hormone (LHRH) agonists and antiandrogens such as: Flutamide, Dutasteride, and Finasteride).
* Subject's Eastern Cooperative Group (ECOG) performance status is 0, 1 or 2 at Screening.
* Subject has acceptable liver function at Screening
* Subject has a normal serum creatinine.
* Subject has acceptable hematologic status at Screening
* Female subjects of childbearing potential (i.e., women who have not been surgically sterilized or have not been post-menopausal for at least one year), and male subjects with partners of childbearing potential, must agree to use medically acceptable methods of contraception beginning on Study Day 1 and continuing until at least four weeks after administration of the subject's final dose of RRx-001.

Exclusion Criteria:

* Impaired cardiac function that in the opinion of the Investigator could interfere with the conduct of the study or could put the subject at unacceptable risk.
* Right-to-left, bidirectional, or transient right-to-left cardiac shunts.
* Subjects with a history of acute cerebral infarction or transient ischemic attack within 90 days prior to Study Day 1.
* Acute myocardial infarction or acute coronary syndromes less than one year prior to enrollment.
* Serious ventricular arrythmias or high risk for arrhythmias due to prolongation of the QT interval.
* Subjects who experienced a major surgery, radiotherapy, or immunotherapy within the last 21 days prior to Study Day 1 (limited palliative radiation is allowed within 14 days prior to Study Day 1).
* Chemotherapy regimens with delayed toxicity within the 28 days prior to Study Day 1 (except for nitrosourea or mitomycin C treatments within 42 days prior to Study Day 1).
* Chemotherapy regimens given continuously or on a weekly basis that Investigator believes to have a limited potential for delayed toxicity within 14 days prior to Study Day 1.
* Use of an investigational anti-cancer drug within 42 days prior to Study Day 1.
* Subject has symptomatic and/or untreated central nervous system metastases and/or intracranial hypertension.
* Subject has a known history of an active and/or an uncontrolled infection with hepatitis A or hepatitis B.
* Subject with a known history of a positive HIV status.
* Subjects with pulmonary edema.
* Subjects with respiratory failure
* Subjects with severe emphysema, pulmonary emboli, pulmonary fibrosis or other conditions that cause pulmonary hypertension due to compromised pulmonary arterial vasculature.
* Subjects with Raynaud's syndrome.
* Subjects with a serious co-morbid medical condition.
* If female, subject is pregnant and/or breastfeeding.
* Any subject with congenital or acquired methemoglobinemia.
* Any subject with a history of inherited anemia or hemoglobinopathy including but not limited to hereditary spherocytosis, hereditary elliptocytosis, hereditary ovalocytosis,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Infante, MD, Principal Investigator — SCRI Development Innovations, LLC; Tony Reid, MD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - Moores University of California San Diego Cancer Center, La Jolla, California
  - Sarah Cannon Research Institute, Nashville, Tennessee

REFERENCES:
- [Derived] Reid T, Oronsky B, Scicinski J, Scribner CL, Knox SJ, Ning S, Peehl DM, Korn R, Stirn M, Carter CA, Oronsky A, Taylor MJ, Fitch WL, Cabrales P, Kim MM, Burris HA Rd, Lao CD, Abrouk NED, Fanger GR, Infante JR. Safety and activity of RRx-001 in patients with advanced cancer: a first-in-human, open-label, dose-escalation phase 1 study. Lancet Oncol. 2015 Sep;16(9):1133-1142. doi: 10.1016/S1470-2045(15)00089-3. Epub 2015 Aug 19. PMID 26296952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Oct 10, 2011, and March 18, 2013, we screened 26 patients from the University of California- San Diego Moores Cancer Center, La Jolla, CA, USA, and the Sarah Cannon Research Institute, Nashville, TN, USA. 25 patients (1 ineligible) were treated.
Pre-assignment Details: One enrolled patient had a disease-associated serious adverse event and died before starting treatment and was not included in the analysis.
Groups:
- RRx-001: Dose Level 1 (10 mg/m2); RRx-001: Dose Level 2 (16.7 mg/m2); RRx-001: Dose Level 3 (24.6 mg/m2); RRx-001: Dose Level 4 (33 mg/m2); RRx-001: Dose Level 5 (55.0 mg/m2); RRx-001: Dose Level 6 (83 mg/m2): Participants received RRx-001 by IV infusion every week for 2 Cycles. On completion, participants were offered further weekly doses, provided the Investigator and Medical Monitor agree it is warranted based on the status and symptomatology of their disease.
Period: Overall Study
Arm/Group | RRx-001: Dose Level 1 (10 mg/m2) | RRx-001: Dose Level 2 (16.7 mg/m2) | RRx-001: Dose Level 3 (24.6 mg/m2) | RRx-001: Dose Level 4 (33 mg/m2) | RRx-001: Dose Level 5 (55.0 mg/m2) | RRx-001: Dose Level 6 (83 mg/m2)
Started | 6 | 3 | 3 | 4 | 3 | 6
Completed | 3 | 3 | 3 | 3 | 3 | 6
Not Completed | 3 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RRx-001: Dose Level 1 (10 mg/m2) | RRx-001: Dose Level 2 (16.7 mg/m2) | RRx-001: Dose Level 3 (24.6 mg/m2) | RRx-001: Dose Level 4 (33 mg/m2) | RRx-001: Dose Level 5 (55.0 mg/m2) | RRx-001: Dose Level 6 (83 mg/m2) | Total
Number analyzed (Participants) | 6 | 3 | 3 | 4 | 3 | 6 | 25
Age, Continuous [Median (Full Range); unit: years] | 59.15 [34.7 to 63.4] | 64.3 [58 to 73.7] | 67.1 [51 to 72.3] | 63.5 [53.8 to 71.1] | 59.5 [57.9 to 70.7] | 58.35 [33.6 to 66.5] | 61.3 [33.6 to 73.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 3 | 2 | 1 | 10
  Male | 5 | 1 | 2 | 1 | 1 | 5 | 15
ECOG Status [Count of Participants; unit: Participants] — Upon enrollment, physicians gave participants an ECOG score of 0-5. (ECOG describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). Lowest score = highest functioning.
  Participants
    ECOG 0 | 2 | 0 | 1 | 1 | 2 | 0 | 6
    ECOG 1 | 3 | 3 | 2 | 3 | 1 | 6 | 18
    ECOG 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Had an Adverse Events
Description: The total number of patients who experienced at least one adverse event while receiving treatment.
Time Frame: From time of receiving a dose of RRx-001 through 92 days
Population: Total number of participants enrolled
Measure: Count of Participants; unit: Participants
Groups:
- RRx-001: Dose Level 1 (10 mg/m2) to Dose Level 5 (83.0 mg/m2): Participants received RRx-001 by IV infusion every week for 2 Cycles. On completion, participants were offered further weekly doses, provided the Investigator and Medical Monitor agree it is warranted based on the status and symptomatology of their disease.
Arm/Group | RRx-001: Dose Level 1 (10 mg/m2) to Dose Level 5 (83.0 mg/m2)
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Arm/Group | RRx-001: Dose Level 1 (10 mg/m2) to Dose Level 5 (83.0 mg/m2)
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 6/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RRx-001: Dose Level 1 (10 mg/m2) to Dose Level 5 (83.0 mg/m2) (N=25)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Emphysematous cholecystitis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RRx-001: Dose Level 1 (10 mg/m2) to Dose Level 5 (83.0 mg/m2) (N=25)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No